CLINICAL TRIAL: NCT06636877
Title: A Randomized, Open-label, Single Dose, Two-way Replicate Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1019" and Co-administration of "BR1019-3" and "BR1019-2" in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1019" and Co-administration of "BR1019-3" and "BR1019-2" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FDC-CT-102
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Essential Hypertension; Type 2 Diabetes
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR1019 (Experimental)
  Interventions: Drug: BR1019
- BR1019-2 + BR1019-3 (Active Comparator)
  Interventions: Drug: BR1019-2; Drug: BR1019-3

INTERVENTIONS:
Drug: BR1019 — One tablet administered alone
  Arms: BR1019
Drug: BR1019-2 — One tablet administered alone
  Arms: BR1019-2 + BR1019-3
Drug: BR1019-3 — One tablet administered alone
  Arms: BR1019-2 + BR1019-3

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and the safety after administration of "BR1019" and co-administration of "BR1019-3" and "BR1019-2" in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those have body mass index (BMI) within the range of 18.0 to 30.0kg/m2 at screening visit.

  * For men, Those who weigh 50 kg or more
  * For women, Those who weigh 45 kg or more
* Those who spontaneously decide to participate and sign written consent to comply with the subject's precautions during the clinical trial period after listening to and fully understanding detailed explanation of this clinical trial
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial*(Except for hormone drugs) from the date of the first administration of the investigational products to 7 days after the last administration and disagrees to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken ETC, OTC, Oriental medicine, health functional food concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetic and pharmacodynamic properties such as Interaction of investigational products, half-life)
* Those who have participated in bioequivalence tests or other clinical trials and administered their investigational products within 6 months prior to the first administration date. (However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal surgery (Except for simple appendectomy, hernia surgery) or gastrointestinal diseases that may affect the absorption of drugs.
* In the case of a female subject, pregnant woman, those suspected pregnancy or lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to time τ | 0-48 hours after administration
Maximum concentration of drug in plasma | 0-48 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No